CLINICAL TRIAL: NCT05187780
Title: Comparison of Spinal Joint Reposition Sense in Idiopathic Scoliosis and Healthy Adolescents
Brief Title: Comparison of Reposition Sense in Scoliosis and Healthy Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Biruni University (Other); Istanbul University (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Asst. Prof., Istanbul University - Cerrahpasa
Other Study IDs: 2020/01
Record Dates: First submitted 2021-12-24; First posted 2022-01-12 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Scoliosis; Adolescence; Healthy; Proprioception
Keywords: scoliosis; proprioception; spine
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Adolescents with Idiopathic Scoliosis who have 10⁰-24⁰ Cobb angles
- Group 2: Adolescents with Idiopathic Scoliosis who have 25⁰-40⁰ Cobb angles
- Group 3: Healthy adolescents without scoliosis as controls

SUMMARY:
The aim of the study is to compare the spine joint reposition sense in adolescent idiopathic scoliosis and healthy adolescents and to investigate whether there is a difference.

DETAILED DESCRIPTION:
Considering the role of proprioception during activities of daily living and exercises, it is important for clinicians and researchers to determine the joint position senses of adolescents with scoliosis and to compare them with their healthy peers in planning appropriate treatment programs. In the light of this information, the aim of the study is to compare the spine joint reposition sense in adolescent idiopathic scoliosis and healthy adolescents and to investigate whether there is a difference. Patients who were diagnosed with Adolescent Idiopathic Scoliosis (AIS) in the Department of Orthopedics and Traumatology of Istanbul University and who were referred to the Department of Physiotherapy and Rehabilitation of the Faculty of Health Sciences of Istanbul University-Cerrahpaşa and Biruni University and their healthy peers will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 10 and 19 years
* Having a Cobb angle of 10-40 degrees measured on the anteroposterior radiograph or a healthy spine alignment (Forward Bend Test < 5⁰ (negative) and Flexicurve Kyphosis Index ≤13)
* No previous conservative approach to scoliosis
* Volunteer to participate in the study

Exclusion Criteria:

* Concomitant mental problem, rheumatological, neuromuscular, cardiovascular, pulmonary history
* Any orthopedic disability or severe pain that would preclude evaluations
* Musculoskeletal injury related to the spine in the last 3 months
* Having had spine surgery
* Presence of tumor in the spine
* Loss of vision and/or hearing/presence of vestibular problems

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents with a diagnosis of idiopathic scoliosis between the ages of 10-19, living in Istanbul and their healthy peers will be included in the study. The subjects will be divided into 3 groups: Group 1: Subjects with AIS with 10⁰-24⁰ Cobb angle, Group 2: Subjects with AIS with 25⁰-40⁰ Cobb angle, Group 3: Healthy adolescents in the same age group (control group).
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2022-01-22 (Actual); Primary Completion 2022-09-22 (Estimated); Study Completion 2022-11-22 (Estimated)

PRIMARY OUTCOMES:
Evaluation of spine joint position reproduction | Baseline
  Acumar™ Dual Inclinometer:
  The subjects will be asked to stay at the reference position for three seconds and then move to the upright position and then go back to the reference angle with their eyes closed. The absolute difference between the two positions in degrees will be noted as the reposition error value. The decrease in the reposition error value is considered as the improvement in the reposition sense.

SECONDARY OUTCOMES:
Spinal pain assessment | Baseline
  Visual Analogue Scale (VAS):
  It is used to quantify the pain intensity of patients. Rest, activity, and night pain will be assessed in the study. The condition that there is no pain is expressed as 0, and the condition that there is too much pain to be tolerated is expressed as 10.
Physical activity level | Baseline
  The subjects' physical activity will be assessed with the Physical Activity Questionnaire for Older Children. The questionnaire consists of a total of 9 items (21 activities) that questions the last 7 days with the form of a 5-point Likert-type. The high scores indicate a high physical activity level. Scoring is based on the frequency of the activities, 'never done' (1 point), '1-2 times' (2 points), '3-4 times' (3 points), '5-6 times' (4 points), ' 7 times and more' (5 points).
Adam's Forward Bending Test | Baseline
  The curve for the diagnosis of scoliosis will be analyzed in the Adam's forward bending test. The test will be performed with a scoliometer to measure the degree of rotation of the vertebrae in the horizontal plane in scoliosis. Rotation measured below 5 degrees is considered normal and does not require follow-up.
Cobb angle assessment | Baseline
  The Cobb method has an important role in determining the size of the spinal curve in frontal plane radiography, determining the size of the treatment, and measuring the effectiveness of the treatment. Cobb angle measurement is performed on standard anteroposterior spine radiography. In the measurement, the angle between a line drawn parallel to the upper vertebra joining the curve and a line drawn parallel to the bottom of the lowest vertebra of the same curve is calculated. The increase in the Cobb degree is considered as an indicator of the increase in the severity of the curvature.
Flexicurve ruler | Baseline
  The ruler, which has a plastic and reshapeable structure, is used for the noninvasive measurement of thoracic kyphosis. The tip of the Flexicurve is placed at C7 and shaped caudally to the contour of the thoracic spine. The Flexicurve is then carefully placed on paper and the outline of the shaped thoracic curve is drawn. This process is repeated three times, straightening the ruler between each measurement. The kyphosis index and Flexicurve angle are calculated using the formulas. The kyphosis index is calculated by dividing the apex of kyphosis by the length of the thoracic curve and multiplying by 100. A kyphosis index value greater than 13 is defined as hyperkyphosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Zengin Aplözgen, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- İstanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)